CLINICAL TRIAL: NCT02991274
Title: A Study of T790M Mutation Testing in Patient Tissue and Blood With Various Detection Platforms at Hospital Laboratories in Comparison With Central Testing
Brief Title: ARTEMIS DIANE T790M (An Amino Acid Substitution at Position 790 in EGFR, From a Threonine (T) to a Methionine (M)) Mutation at Hospital Laboratories in Comparison With Central Laboratory
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160C00041
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Locally Advanced or Metastatic EGFR(+) NSCLC Patients
Keywords: T790M; EGFR (Epidermal Growth Factor Receptor) mutation; NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T790M mutation test: genomic testing of T790M mutation
  Interventions: Procedure: genomic testing of T790M mutation

INTERVENTIONS:
Procedure: genomic testing of T790M mutation — patients will need to have genomic testing of T790M mutation at hospital laboratories and in central laboratory.

SUMMARY:
The study primary objective is to assess the concordance of T790M resistance mutation testing from hospital-based laboratories with T790M resistance mutation testing from a central laboratory.

DETAILED DESCRIPTION:
This is a multi-center testing study. 800 patients from 80 different hospital sites will have local T790M testing by different molecular testing platforms and have central testing by Cobas platform. These two sets of data (local T790M testing and central T790M testing) will be analysed and compared to assess the concordance of these T790M testing platforms.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent or EC approve informed consent waiver prior to any study specific procedures
2. Histological or cytological confirmed locally advanced NSCLC (stage IIIB) or metastatic (stage IV) NSCLC, not amenable to curative surgery or radiotherapy.
3. Patients who have progressed following prior therapy with an EGFR-TKI agent.
4. Patients who consent to provide tumour tissue and/or blood.

Exclusion Criteria:

1. Patients who disagree to participate this study.
2. Patients whose medical objection was recorded to use the existing data from medical practice for scientific research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 897 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
the concordance of T790M mutation testing between the test in central and local labs | within 1 -14 days after enrolled
  Concordance (%)=(number of patients with same T790M mutation status based on central and local labs)/(total number of patients in the FAS) ×100%

SECONDARY OUTCOMES:
The prevalence rate of T790M mutation based on the central lab testing | within 1 -14 days after enrolled
  Prevalence (%) = (number of patients with T790M mutation positive)/(total number of patients in the FAS)×100%
The sensitivity of each platform based on the local lab plasma testing | within 1 -14 days after enrolled
  Sensitivity (%)=(number of patients with T790M mutation positive based on both tissue and plasma tests)/(number of patients with T790M mutation positive based on tissue test) ×100%
The Specificity of each platform based on the local lab plasma testing | within 1 -14 days after enrolled
  Specificity (%)=(number of patients with T790M mutation negative based on both tissue and plasma tests)/(number of patients with T790M mutation negative based on tissue test) ×100%
The Positive predictive value of each platform based on the local lab plasma testing | within 1 -14 days after enrolled
  Positive predictive value (%)=(number of patients with T790M mutation positive based on both tissue and plasma tests)/(number of patients with T790M mutation positive based on plasma test) ×100%
The Negative predictive value of each platform based on the local lab plasma testing | within 1 -14 days after enrolled
  Negative predictive value (%)=(number of patients with T790M mutation negative based on both tissue and plasma tests)/(number of patients with T790M mutation negative based on plasma test) ×100%
The Concordance of each platform based on the local lab testing | within 1 -14 days after enrolled
  Concordance (%)=(number of patients with same T790M mutation status based on tissue and plasma tests)/(total number of patients in the FAS) ×100%
The prevalence of C797S (An amino acid substitution at position 797 in EGFR, from a Cysteine (C) to a Serine (S) ) resistance mutation based on the local lab testing | within 1 -14 days after enrolled
  Prevalence (%) = (number of patients with C797S mutation positive)/(total number of patients with evaluable C797S testing)×100%
Rare EGFR mutation prevalence rate | within 1-14 days after enrolled
  Prevalence (%) = (number of patients with rare EGFR mutation positive)/(total number of patients in the FAS)×100%

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Jie He, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jie Wang, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (22):
- China (22):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yantai
  - Research Site, Zhengzhou